CLINICAL TRIAL: NCT06119165
Title: Impact of Environmental Nudges on Dietary Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-1785
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-10

CONDITIONS: Healthy Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will conduct online shopping tasks without any environmental nudges. This includes no labels, peer comparison messages, or suggested product swaps.
- Environmental (Experimental): Participants in the experimental arm will shop and receive environmental nudges in the form of labels, peer comparisons messages, and suggested product swaps.
  Interventions: Behavioral: Environmental nudges

INTERVENTIONS:
Behavioral: Environmental nudges — Participants will view protein, frozen meal, and snack products with eco-labels applied. For each category, they will then be instructed to select 1 item from that category they wish most to purchase. Categories will be shown in random order. If a participant selects a product with a red eco-label, they will be shown a peer comparison message and will be given an opportunity to switch to a product with a yellow or green eco-label.
  Arms: Environmental

SUMMARY:
Purpose: The overall purpose of this study is to evaluate the impact of a suite of environmentally focused nudges on the nutritional quality of consumers' food selections.

Participants: ~2,000 US adults ages 18-25, at least 25% currently enrolled full-time in college, recruited from CloudResearch Prime Panels.

Procedures: Participants will be randomly assigned to view food products with or without environmental nudges (eco-labels, peer comparison message, and swaps). They will be asked to select items that they most wish to purchase and will then be asked a series of questions about the products and nudges. Questions will also include standard socio-demographic variables.

DETAILED DESCRIPTION:
Participants will be recruited from CloudResearch Prime Panels (an online panel research company). Study participants include 2,000 young adults between 18 and 25 years old with at least 25% currently enrolled in college, recruited to match census distribution of race/ethnicity and gender. Participants will electronically acknowledge their consent to participate in the study.

On the study platform (Qualtrics), participants will be randomly assigned to 1 of 2 arms with equal probability. Participants will complete a shopping task via an online 9-minute survey. They will view products displayed as if they were offered from a grocery store. Products will be frozen meals, such as burritos and pizza, snack items such as dried fruit and chips, and protein items, such as ground beef and chicken breasts. They will then be instructed to select 1 item they most wish to purchase from each category.

Participants in the experimental arm will shop and receive environmental nudges in the form of labels, feedback, peer comparisons, and suggested product swaps. In the control arm, participants will conduct online shopping tasks without any environmental nudges. After selecting products, participants will answer questions about the products and labels, as well as standard socio-demographic questions.

ELIGIBILITY:
Inclusion criteria:

* 18 to 25 years old
* Currently resides in the United States

Exclusion criteria:

* Completion of the survey in <1/3 of the median completion time

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2132 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Nutri-Score Scores | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Healthfulness of product selections (operationalized as products' Nutri-Score scores). Products' Nutri-Score scores are calculated using the updated 2022 algorithm released by the Scientific Committee of the Nutri-Score (ScC). Scores range from -15 (Nutri-Score of "A") to 40 (Nutri-Score of "E"), with lower scores indicating a more healthful product selection.

SECONDARY OUTCOMES:
Carbon Footprint | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Carbon footprint of product selections [operationalized as products' greenhouse gas emissions (GHGE) per 100g].
Acceptability of Eco-Label Intervention | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Acceptability of eco-labels on products, measured by an item adapted from Vargas-Meza et al., 2019. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "A great deal" (coded as 5), with higher scores representing a higher acceptability of eco-labels.
Acceptability of Swaps Intervention | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Acceptability of environmental swaps, measured by an item adapted from Vargas-Meza et al., 2019. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "A great deal" (coded as 5), with higher scores representing a higher acceptability of swaps.
Acceptability of Peer Comparison Message Intervention | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Acceptability of peer comparison messages, measured by an item adapted from Vargas-Meza et al., 2019. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "A great deal" (coded as 5), with higher scores representing a higher acceptability of peer comparison messages.
Health Elaboration | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  How much the participant reports thinking about the healthfulness of products when making selections. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "A great deal" (coded as 5), with higher scores representing a higher amount of thinking about the healthfulness of products.
Taste Elaboration | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  How much the participant reports thinking about the taste of products when making selections. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "A great deal" (coded as 5), with higher scores representing a higher amount of thinking about the taste of products.
Cost Elaboration | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  How much the participant reports thinking about the cost of products when making selections. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "A great deal" (coded as 5), with higher scores representing a higher amount of thinking about the cost of products.
Environmental Sustainability Elaboration | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  How much the participant reports thinking about the environmental sustainability of products when making selections. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "A great deal" (coded as 5), with higher scores representing a higher amount of thinking about the environmental sustainability of products.
Perceived Healthfulness of Sustainable Products | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' perceptions about the healthfulness of sustainable products. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "Extremely" (coded as 5), with higher scores representing a higher perceived healthfulness of sustainable products.
Perceived Healthfulness of Unsustainable Products | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' perceptions about the healthfulness of unsustainable products. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "Extremely" (coded as 5), with higher scores representing a higher perceived healthfulness of unsustainable products.
Perceived Sustainability of Sustainable Products | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' perceptions about the sustainability of sustainable products. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "Extremely" (coded as 5), with higher scores representing a higher perceived sustainability of sustainable products.
Perceived Sustainability of Unsustainable Products | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' perceptions about the sustainability of unsustainable products. Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "Extremely" (coded as 5), with higher scores representing a higher perceived sustainability of unsustainable products.
Purchase Intentions of Sustainable Products | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' intentions to purchase a sustainable product in the next month. Likert responses are on a 1 to 5 scale, from "Not at all likely" (coded as 1) to "Extremely likely" (coded as 5), with higher scores representing a higher intention to purchase.
Purchase Intentions of Unsustainable Products | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' intentions to purchase an unsustainable product in the next month. Likert responses are on a 1 to 5 scale, from "Not at all likely" (coded as 1) to "Extremely likely" (coded as 5), with higher scores representing a higher intention to purchase.
Injunctive Norms | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' perceived approval from people important in their life for purchasing environmentally sustainable products. Likert responses are on a 1 to 5 scale, from "Strongly disagree" (coded as 1) to "Strongly agree" (coded as 5), with higher scores representing higher perceived approval about purchasing environmentally sustainable products.
Descriptive Norms | Immediately after exposure to intervention and product selection task, assessed during 1-time online study visit
  Participants' belief that most shoppers purchase environmentally sustainable foods when shopping for groceries. Likert responses are on a 1 to 5 scale, from "Strongly disagree" (coded as 1) to "Strongly agree" (coded as 5), with higher scores representing higher belief that most shoppers purchase environmentally sustainable foods.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Smith Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Anna H Grummon, PhD, Principal Investigator — Stanford University
Locations (1):
- UNC Carolina Population Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset and the corresponding survey codebook will be published to a data repository. The study protocol, statistical analysis plan, and informed consent form will be published alongside as supplementary material.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The deidentified dataset and corresponding survey codebook will be available upon publication of study results and will be available indefinitely.
Access Criteria: Anyone who wishes to access the data.

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT06119165/SAP_000.pdf